CLINICAL TRIAL: NCT01807585
Title: VenaSeal Sapheon Closure System vs. Radiofrequency Ablation for Incompetent Greater Saphenous Veins
Brief Title: VenaSeal Sapheon Closure System Pivotal Study (VeClose)
Acronym: VeClose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Collaborators: Sapheon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-11101-01
Record Dates: First submitted 2013-03-05; First posted 2013-03-08 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Great Saphenous Vein (GSV) With Venous Reflux Disease
Keywords: GSV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VenaSeal SCS (Experimental): Endovenous delivery of VenaSeal Adhesive (VA) to a target site in diseased great saphenous veins (GSV). The VA is dispensed in small amounts with each pull of the trigger equaling 0.10 cc. Subjects were randomized in a 1:1 ratio to either VenaSeal SCS or to RFA.
  Interventions: Device: VenaSeal SCS
- RFA (ClosureFast) (Active Comparator): Endovenous insertion of the ClosureFast radiofrequency ablation (RFA) catheter into a target site in diseased great saphenous veins (GSV). Heat is applied to the target vein using radiofrequency energy to ablate the target vein. Subjects were randomized in a 1:1 ratio to either VenaSeal SCS or RFA.
  Interventions: Device: ClosureFast Radiofrequency Ablation (RFA)
- Roll-in (VenaSeal SCS) (Experimental): Prior to initiation of the randomized cohort at each site, a non-randomized cohort of 2 subjects per clinical site (roll-in phase) were enrolled and treated with VenalSeal SCS with endovenous delivery of VenaSeal Adhesive (VA) to a target site in diseased great saphenous veins (GSV). The VA is dispensed in small amounts with each pull of the trigger equaling 0.10 cc.
  Interventions: Device: Roll-in (VenaSeal SCS)

INTERVENTIONS:
Device: VenaSeal SCS — Non-tumescent, non-thermal, non-sclerosant procedure that uses a proprietary medical adhesive delivered endovenously to close the vein.
  Other Names: VenaSeal Sapheon Closure System; VSCS
  Arms: VenaSeal SCS
Device: ClosureFast Radiofrequency Ablation (RFA) — Radiofrequency thermal ablation of the GSV using the Covidien ClosureFast system.
  Other Names: ClosureFast
  Arms: RFA (ClosureFast)
Device: Roll-in (VenaSeal SCS) — Non-tumescent, non-thermal, non-sclerosant procedure that uses a proprietary medical adhesive delivered endovenously to close the vein.
  Other Names: VenaSeal Sapheon Closure System; VSCS; Roll-in
  Arms: Roll-in (VenaSeal SCS)

SUMMARY:
The VeClose pivotal study was a controlled, randomized, prospective, multicenter, pivotal study in which patients with venous reflux in the great saphenous vein (GSV) were treated with either the VenaSeal closure system (VenaSeal SCS) or radiofrequency ablation (RFA) therapy.

DETAILED DESCRIPTION:
The purpose of the VeClose study was to demonstrate safety and effectiveness of the VenaSeal SCS as being both 1) non-inferior to RFA therapy in achieving anatomical closure of lower extremity superficial truncal veins in patients with venous reflux through endovascular transcatheter embolization with coaptation of the GSV at 3 months, and 2) superior in the reduction of intraprocedural and post procedural pain and symptoms as compared to treatment with RFA.

The study was designed to demonstrate safety of the VenaSeal SCS by follow-up visits that evaluated, via duplex ultrasound and physical exam, the presence of deep vein thrombosis and/or pulmonary embolus.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years and ≤ 70 years of age at the time of screening
2. Reflux in the great saphenous vein (GSV) greater than 0.5 sec reflux
3. One or more of the following symptoms related to the target vein: aching, throbbing, heaviness, fatigue, pruritis, night cramps, restlessness, generalized pain or discomfort, swelling
4. GSV diameter while standing of 3-12 mm throughout the target vein as measured by Duplex ultrasound
5. Clinical, etiology, assessment and pathophysiology (CEAP) classification of C2 (if symptomatic) - C4b
6. Ability to walk unassisted
7. Ability to attend follow-up visits
8. Ability to understand the requirements of the study and to provide informed consent

Exclusion Criteria:

1. Life expectancy < 1 year
2. Active treatment for malignancy other than non-melanoma skin cancer
3. Symptomatic peripheral arterial disease with ankle-brachial index (ABI) <0.89
4. Daily use of narcotic or non-steroidal anti-inflammatory pain medications to control pain associated with GSV reflux
5. Current, regular use of systemic anticoagulation (e.g., warfarin, heparin)
6. Previous or suspected deep vein thrombosis (DVT) or pulmonary embolus (PE)
7. Previous superficial thrombophlebitis in GSV
8. Previous treatment of venous disease in target limb, other than spider vein treatment
9. Known hypercoagulable disorder
10. Conditions which prevent vein treatment with either RFA or VenaSeal SCS
11. Immobilization or inability to ambulate
12. Pregnant prior to enrollment
13. Tortuous GSV, which, in the opinion of the investigator, will limit catheter placement or require more than one primary access site
14. Aneurysm of the target vein with local diameter >12 mm
15. Significant, incompetent, ipsilateral small saphenous, intersaphenous or anterior accessory great saphenous vein(s)
16. Known sensitivity to cyanoacrylate (CA) adhesives
17. Current participation in another clinical study involving an investigational agent or treatment, or within the 30 days prior to enrollment
18. Patients who require bilateral treatment during the next 3 months
19. Patients who require additional ipsilateral treatments on the same leg within 3 months following treatment

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Morrison, MD, Principal Investigator — Morrison Vein Institute
Locations (10):
- United States (10):
  - Morrison Vein Institute, Scottsdale, Arizona
  - GBK Cosmetic Laser Dermatology, San Diego, California
  - Radiology Imaging Associates (RIA), Greenwood Village, Colorado
  - Vein Clinics of America, Oakbrook Terrace, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - MD Laser Skin & Vein Institute, Hunt Valley, Maryland
  - Vein Institute of Buffalo, North Tonawanda, New York
  - Inovia Vein Specialty Center, Bend, Oregon
  - Sentara Vascular Specialist, Virginia Beach, Virginia
  - Lake Washington Vascular, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morrison N, Gibson K, Vasquez M, Weiss R, Cher D, Madsen M, Jones A. VeClose trial 12-month outcomes of cyanoacrylate closure versus radiofrequency ablation for incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2017 May;5(3):321-330. doi: 10.1016/j.jvsv.2016.12.005. Epub 2017 Mar 6. PMID 28411697
- [Result] Kolluri R, Gibson K, Cher D, Madsen M, Weiss R, Morrison N. Roll-in phase analysis of clinical study of cyanoacrylate closure for incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2016 Oct;4(4):407-15. doi: 10.1016/j.jvsv.2016.06.017. Epub 2016 Aug 8. PMID 27638993
- [Derived] Gibson K, Morrison N, Kolluri R, Vasquez M, Weiss R, Cher D, Madsen M, Jones A. Twenty-four month results from a randomized trial of cyanoacrylate closure versus radiofrequency ablation for the treatment of incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2018 Sep;6(5):606-613. doi: 10.1016/j.jvsv.2018.04.009. Epub 2018 Jun 15. PMID 29914814
- [Derived] Morrison N, Gibson K, McEnroe S, Goldman M, King T, Weiss R, Cher D, Jones A. Randomized trial comparing cyanoacrylate embolization and radiofrequency ablation for incompetent great saphenous veins (VeClose). J Vasc Surg. 2015 Apr;61(4):985-94. doi: 10.1016/j.jvs.2014.11.071. Epub 2015 Jan 31. PMID 25650040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The VeClose pivotal study was a prospective, multicenter, randomized, controlled study in which patients with venous reflux in the great saphenous vein (GSV) were treated with either VenaSeal SCS or radiofrequency ablation (RFA) therapy. Patients were treated between March 2013 and September 2013. There were 10 sites with 242 subjects.
Pre-assignment Details: The VeClose study had two phases: a roll-in phase and a randomization phase. At each site, the first two enrolled subjects were treated with VenaSeal SCS only (no randomization) as "roll-in cases". Following completion of the roll-in phase, the site entered the randomized phase where subjects were assigned to either VenaSeal SCS or RFA cohort.
Groups:
- Roll-In (VenaSeal SCS): Endovenous delivery of VenaSeal Adhesive (VA) to a target site in diseased great saphenous veins (GSV). At each site, the first two enrolled subjects were treated with VenaSeal SCS only (no randomization). These subjects underwent the same preoperative and postoperative assessments (with the same schedule) as patients who underwent randomization.
- VenaSeal SCS (Randomized Phase): Endovenous delivery of VenaSeal Adhesive (VA) to a target site in diseased great saphenous veins (GSV). Following completion of the Roll-in phase, subjects were then randomized at each site in a 1:1 fashion to either VenaSeal SCS or RFA.
- RFA (Randomized Phase): Endovenous insertion of the ClosureFast radiofrequency ablation (RFA) catheter into a target site in diseased great saphenous veins (GSV). Following completion of the Roll-in phase, subjects were then randomized at each site in a 1:1 fashion to either VenaSeal SCS or RFA.
Period: Overall Study
Arm/Group | Roll-In (VenaSeal SCS) | VenaSeal SCS (Randomized Phase) | RFA (Randomized Phase)
Started (Date of first Baseline Visit) | 20 | 108 | 114
3 Mos (Primary endpoint) | 20 | 108 | 113
Completed | 19 | 104 | 108
Not Completed | 1 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roll-In (VenaSeal SCS) | VenaSeal SCS (Randomized Phase) | RFA (Randomized Phase) | Total
Number analyzed (Participants) | 20 | 108 | 114 | 242
Age, Continuous [Mean (Full Range); unit: years] | 53.1 [36 to 65] | 49.0 [26 to 70] | 50.5 [25 to 70] | 50.1 [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 83 | 93 | 193
  Male | 3 | 25 | 21 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Closure of the Target Vein at 3 Months
Description: The primary endpoint of the study was complete closure of the target vein at 3 months after index treatment as judged by the vascular ultrasound laboratory. Complete closure was defined as Doppler ultrasound examination showing closure along the entire treated vein segment with no discrete segments of patency exceeding 5 cm.
Time Frame: 3 months
Population: Primary effectiveness was analyzed on the randomized cohort only and used an Intent to Treat (ITT) population, consisting of all treated subjects. The difference in success rates was calculated after imputing missing values with various methods.
Measure: Count of Participants; unit: Participants
Arm/Group | VenaSeal SCS (Randomized Phase) | RFA (Randomized Phase)
Number analyzed (Participants) | 108 | 114
Participants | 107 | 109
Statistical Analysis 1: Comparison: VenaSeal SCS (Randomized Phase) vs RFA (Randomized Phase); Last Observation Carried Forward (LOCF); Test type: Non-Inferiority — Non-inferiority was determined by the application of a Z-test with a 10% non-inferiority margin as well as examination of confidence intervals; p < 0.0001, One tailed Z-test; Risk Difference (RD) = 3.5, 95% CI 2-sided [-0.7 to 7.6]

2. Secondary Outcome: Intraoperative Pain
Description: After the procedure, pain experienced during the procedure was rated by the subjects on a 0-10 numeric rating scale (NRS) where 0 represents no pain whatsoever and 10 represents worst imaginable pain.
Time Frame: During the operative procedure, which was an average of 24 minutes for VenaSeal SCS, 19 minutes for RFA, and 31 minutes for Roll-in group.
Population: Completed Case (CC) analysis population consisted of all treated subjects for whom data were available for the endpoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Roll-In (VenaSeal SCS) | VenaSeal SCS (Randomized Phase) | RFA (Randomized Phase)
Number analyzed (Participants) | 18 | 106 | 113
scores on a scale | 1.28 (1.53) | 2.16 (2.23) | 2.35 (2.18)

3. Secondary Outcome: Ecchymosis at Day 3
Description: At the Day 3 visit, the investigator visually rated the subject's ipsilateral leg for the occurrence of ecchymosis along the treated area based on a Scale for Ecchymosis Assessment with a 0-5 rating scale, with 0 being the best possible outcome and 5 being the worst possible outcome.
  The treatment area was defined as the area of skin overlying the treated vein, excluding the 5 cm of skin immediately adjacent to the access site.
  The rating scale was based on the percentage of ecchymosis of the treated area according to the following criteria:
  0 rating = no ecchymosis,
  1. rating = less than 25% ecchymosis,
  2. rating = 25-50% ecchymosis,
  3. rating = 50-75% ecchymosis,
  4. rating = 75-100% ecchymosis,
  5. rating = extension of ecchymosis above or below the treated area.
Time Frame: First follow up visit at day 3
Population: Completed Case (CC) analysis population consisted of all treated subjects for whom data were available for the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Roll-In (VenaSeal SCS) | VenaSeal SCS (Randomized Phase) | RFA (Randomized Phase)
Number analyzed (Participants) | 20 | 108 | 114
Participants
  None | 15 | 73 | 55
  <25% | 5 | 29 | 38
  25-50% | 0 | 3 | 16
  50-75% | 0 | 2 | 4
  75-100% | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Roll-In (VenaSeal SCS) | VenaSeal SCS (Randomized Phase) | RFA (Randomized Phase)
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/108 | 0/114
Serious Adverse Events (participants affected / at risk) | 1/20 | 5/108 | 6/114
Other Adverse Events (participants affected / at risk) | 7/20 | 26/108 | 15/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roll-In (VenaSeal SCS) (N=20) | VenaSeal SCS (Randomized Phase) (N=108) | RFA (Randomized Phase) (N=114)
Ischemic Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Symptomatic orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Left hip bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Left knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Liver cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non ST elevation MI (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Right breast invasive lobular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Right knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roll-In (VenaSeal SCS) (N=20) | VenaSeal SCS (Randomized Phase) (N=108) | RFA (Randomized Phase) (N=114)
Phlebitis in treatment zone (Vascular disorders) | 2 (2) | 12 (13) | 9 (9)
Phlebitis not in treatment zone (Vascular disorders) | 0 (0) | 8 (8) | 6 (6)
Superficial vein thrombophlebitis (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Other (Musculoskeletal and connective tissue disorders) | 2 (3) | 8 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No